CLINICAL TRIAL: NCT00173459
Title: Dynamic Profiles of Cytokine/Chemokine in Severe Acute Respiratory Syndrome
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700671
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-07

CONDITIONS: SARS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Severe acute respiratory syndrome (SARS) is an emerging infectious disease caused by a novel coronavirus (SARS-CoV). The major clinical features of SARS include fever, dyspnea, lymphopenia, and a rapid progression of pulmonary infiltrates on chest radiologic images. The SARS-related deaths have resulted mainly from pulmonary complications, including progressive respiratory failure due to alveolar damage and acute respiratory distress syndrome (ARDS). Pathological changes in SARS suggest that SARS sequelae such as infiltration of PMN in lung tissue, multiple organ dysfunction and ARDS have been associated with cytokines and chemokine dysregulation. Some patients still manifested lung injury at a time when the viral load was falling also supports the immune nature of the lung damage. We therefore undertook an analysis of dynamic production of cytokine/chemokines in SARS patients with an initial normal chest radiograph in order to improve understanding of disease pathogenesis and improve patient management.

ELIGIBILITY:
Inclusion Criteria:

* SARS group: Patients with SARS

Exclusion Criteria:

* Hospital acquired pneumonia

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yien Chien, MD, Study Chair — NTUH